CLINICAL TRIAL: NCT00404092
Title: A Phase II Dose Escalation Study of Caspofungin in Patients With Invasive Aspergillosis
Brief Title: Caspofungin Maximum Tolerated Dose in Patients With Invasive Aspergillosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Oliver Cornely, MD, Prof. Dr. Oliver Cornely, University of Cologne
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln-687; 2006-001936-30 (EudraCT Number)
Record Dates: First submitted 2006-11-24; First posted 2006-11-27 (Estimated); Results first posted 2013-01-21 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Invasive Aspergillosis
Keywords: aspergillosis; caspofungin; maximum tolerated dose
MeSH Terms: conditions — Aspergillosis | interventions — Caspofungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1st cohort (Experimental): 70mg caspofungin 1x/day
  Interventions: Drug: caspofungin
- 2nd cohort (Experimental): 100mg caspofungin 1x/day
  Interventions: Drug: caspofungin
- 3rd cohort (Experimental): 150mg caspofungin 1x/day
  Interventions: Drug: caspofungin
- 4th cohort (Experimental): 200mg caspofungin 1x/day
  Interventions: Drug: caspofungin

INTERVENTIONS:
Drug: caspofungin — i.v.
  Other Names: cancidas

SUMMARY:
This study investigates the safety and tolerability as well as the efficacy and pharmacokinetics of caspofungin in four escalating dosages in adult patients with hematologic malignancies and proven or probable invasive aspergillosis.

DETAILED DESCRIPTION:
Due to its efficacy and a broad antifungal spectrum against relevant fungal pathogens, lack of cross-resistance to azoles and amphotericin B, documented efficacy against human Aspergillus infections, favorable pharmacokinetic properties, and excellent tolerability according to the current data, caspofungin is a highly promising candidate for improving the results of treatment of invasive fungal infections.

Preclinical and clinical data indicate a dose dependent antifungal efficacy of caspofungin as well as of other echinocandins such as micafungin and anidulafungin. Thus it appears reasonable to investigate the impact of higher doses of caspofungin to improve the results already achieved with this component so far.

The maximum tolerated dose (MTD) of caspofungin and the distribution of the drug in patients following administration of doses of 70 mg or more are not yet known. We therefore investigate the safety, tolerability and pharmacokinetics of caspofungin in rising doses in a dose escalation study in adult patients with proven or probable invasive aspergillosis.

ELIGIBILITY:
Inclusion Criteria:

* Immunocompromised due to hematologic malignancies, bone marrow failure syndromes, hematopoietic stem cell transplantation, solid organ transplantation, other conditions resulting in severe neutropenia, HIV infection, prolonged corticosteroid therapy, treatment with other immunosuppressive medications, or other immunocompromising conditions that place patients at risk for invasive fungal infections.
* Evidence of proven or probable invasive aspergillosis, by modified EORTC criteria

Exclusion Criteria:

* Concomitant other systemic antifungal agents are not permitted on study.
* Chronic invasive fungal infection, defined as signs/symptoms of invasive fungal infection present for > 4 weeks preceding entry into study
* Prior systemic therapy of ≥ 4 days with any polyene anti-fungal agent within 14 days of study enrollment
* Prior systemic therapy of ≥ 4 days with non-polyenes for the current, documented IFI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2006-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver A. Cornely, MD, Principal Investigator — Klinikum der Universität zu Köln
Locations (4):
- University Hospital Gasthuisberg, Leuven, Belgium
- Germany (3):
  - Charité - Campus Benjamin Franklin, Berlin
  - Klinikum der Universität zu Köln, Cologne
  - Universitätsklinikum Münster, Münster

REFERENCES:
- [Result] Cornely OA, Vehreschild JJ, Vehreschild MJ, Wurthwein G, Arenz D, Schwartz S, Heussel CP, Silling G, Mahne M, Franklin J, Harnischmacher U, Wilkens A, Farowski F, Karthaus M, Lehrnbecher T, Ullmann AJ, Hallek M, Groll AH. Phase II dose escalation study of caspofungin for invasive Aspergillosis. Antimicrob Agents Chemother. 2011 Dec;55(12):5798-803. doi: 10.1128/AAC.05134-11. Epub 2011 Sep 12. PMID 21911573
- [Result] Wurthwein G, Cornely OA, Trame MN, Vehreschild JJ, Vehreschild MJ, Farowski F, Muller C, Boos J, Hempel G, Hallek M, Groll AH. Population pharmacokinetics of escalating doses of caspofungin in a phase II study of patients with invasive aspergillosis. Antimicrob Agents Chemother. 2013 Apr;57(4):1664-71. doi: 10.1128/AAC.01912-12. Epub 2013 Jan 18. PMID 23335740

RESULTS

PARTICIPANT FLOW:
Groups:
- 1st Cohort: 70mg 1x/day
  caspofungin : i.v.
- 2nd Cohort: 100mg 1x/day
  caspofungin : i.v.
- 3rd Cohort: 150mg 1x/day
  caspofungin : i.v.
- 4th Cohort: 200mg 1x/day
  caspofungin : i.v.
Period: Overall Study
Arm/Group | 1st Cohort | 2nd Cohort | 3rd Cohort | 4th Cohort
Started | 9 | 8 | 9 | 20
Completed | 8 | 8 | 8 | 20
Not Completed | 1 | 0 | 1 | 0
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1st Cohort | 2nd Cohort | 3rd Cohort | 4th Cohort | Total
Number analyzed (Participants) | 9 | 8 | 9 | 20 | 46
Age, Customized [Number; unit: participants]
  <=30 years | 0 | 1 | 0 | 1 | 2
  Between 30 and 40 years | 2 | 1 | 1 | 2 | 6
  Between 40 and 50 years | 1 | 1 | 2 | 2 | 6
  Between 50 and 60 years | 3 | 0 | 1 | 3 | 7
  Between 60 and 70 years | 2 | 4 | 4 | 7 | 17
  > 70 years | 1 | 1 | 1 | 5 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 4 | 10 | 21
  Male | 7 | 3 | 5 | 10 | 25
Region of Enrollment [Number; unit: participants]
  Germany | 9 | 8 | 9 | 20 | 46

OUTCOME MEASURES:

1. Secondary Outcome: Efficacy of Caspofungin in Four Escalating Dosages in the Treatment of Proven or Probable Invasive Aspergillosis.
Description: Numbers of patients in each dose cohort according to invasive aspergillosis (IA) outcome at end of protocol treatment (EOT), 4 weeks follow-up (4w FU) and 12 weeks follow-up (12w FU), respectively. 12w FU was only required for patients with a CR or PR at the 4w FU.
  Definitions:
  CR: resolution of all attributable symptoms, signs, and radiographic or bronchoscopic abnormalities.
  PR: clinically meaningful improvement in attributable symptoms, signs, and radiographic (min. 50% decrease) or bronchoscopic abnormalities.
  Stable disease (SD): no improvement in attributable symptoms, signs, and radiographic or bronchoscopic abnormalities.
  Failure: deterioration in attributable clinical or radiographic abnormalities necessitating alternative antifungal therapy or resulting in death.
  Relapse: reemergence of IA after EOT following CR, PR or SD or early withdrawal.
Time Frame: End of caspofungin treatment; 4 weeks follow-up; 12 weeks follow-up
Population: All 46 recruited patients were included in the analysis. 2 (EOT), 16 (4w FU) and 23 (12w FU) outcomes out of 46 were not recorded.
Measure: Number; unit: participants
Arm/Group | 1st Cohort | 2nd Cohort | 3rd Cohort | 4th Cohort
Number analyzed (Participants) | 9 | 8 | 9 | 20
participants
  Favorable Response (CR&PR) | 4 | 3 | 6 | 12
  Complete Response (CR) | 0 | 0 | 1 | 0
  Partial Response (PR) | 4 | 3 | 5 | 12
  Stable Disease | 2 | 0 | 2 | 0
  Failure | 3 | 4 | 0 | 8
  Relapse (from Favorable Response) 4w post EOT | 0 | 0 | 2 | 3
  Relapse (from Favorable Response) 12w post EOT | 1 | 0 | 2 | 3

2. Primary Outcome: Safety and Tolerability of Caspofungin in Four Escalating Dosages in Adult Patients With Hematologic Malignancies and Proven or Probable Invasive Aspergillosis
Description: Endpoints of safety and tolerability are the number of toxicity-related study therapy discontinuations and grade III and IV clinical and laboratory events, as evaluated on the basis of current NCI criteria.
Time Frame: End of caspofungin treatment, treatment duration varied between 3 and 29 days (mean: 20.5; median: 24.5)
Measure: Number; unit: events
Arm/Group | 1st Cohort | 2nd Cohort | 3rd Cohort | 4th Cohort
Number analyzed (Participants) | 9 | 7 | 8 | 20
events
  Treatment-emergent AEs (grade 3 to 5) | 11 | 12 | 9 | 73
  At least possibly related AEs (grade 3 to 5) | 0 | 0 | 0 | 6
  At least probably related AEs (grade 3 to 5) | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Arm/Group | 1st Cohort | 2nd Cohort | 3rd Cohort | 4th Cohort
Serious Adverse Events (participants affected / at risk) | 1/9 | 5/8 | 7/9 | 12/20
Other Adverse Events (participants affected / at risk) | 9/9 | 8/8 | 9/9 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1st Cohort (N=9) | 2nd Cohort (N=8) | 3rd Cohort (N=9) | 4th Cohort (N=20)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Psychosis (Psychiatric disorders) | 0 | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Hypotension (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Syncope (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 3
Liver failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 3
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Fever (General disorders) | 0 | 0 | 4 | 3
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Worsening of general condition (General disorders) | 0 | 1 | 0 | 0
Death (General disorders) | 1 | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Persistence or progression of underlying disease (General disorders) | 0 | 0 | 1 | 4
Urinary bladder tamponade (Surgical and medical procedures) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1st Cohort (N=9) | 2nd Cohort (N=8) | 3rd Cohort (N=9) | 4th Cohort (N=20)
intermittant ear pressure (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
pressure on the ears (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 11
intermittend leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
intermittend thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0
persistence of blast cells (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
persistence of blasts (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
thrombopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 3
arterial hypertension (Cardiac disorders) | 0 | 0 | 0 | 1
cardiac dysrrhthmias (Cardiac disorders) | 0 | 0 | 0 | 1
circulatory discomfort (Cardiac disorders) | 0 | 1 | 0 | 0
collaps (Cardiac disorders) | 0 | 1 | 0 | 1
cyanosis (Cardiac disorders) | 0 | 1 | 0 | 0
edema (Cardiac disorders) | 5 | 1 | 2 | 4
fall, knocked head (Cardiac disorders) | 1 | 0 | 0 | 0
heart-trouble (Cardiac disorders) | 1 | 0 | 0 | 0
hypertension (Cardiac disorders) | 0 | 1 | 0 | 3
hypotension (Cardiac disorders) | 2 | 0 | 0 | 1
hypotension with dizziness (Cardiac disorders) | 0 | 0 | 0 | 1
hypotonia (Cardiac disorders) | 1 | 0 | 0 | 0
tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0
tightness in the chest (Cardiac disorders) | 0 | 1 | 1 | 0
vertigo (Cardiac disorders) | 1 | 1 | 2 | 1
thrombosis left leg (Vascular disorders) | 0 | 1 | 0 | 0
fatigue (General disorders) | 0 | 0 | 1 | 0
fatique (General disorders) | 0 | 1 | 0 | 1
loss of weight (General disorders) | 1 | 0 | 0 | 0
night sweat (General disorders) | 0 | 0 | 0 | 2
perspiration (General disorders) | 0 | 0 | 0 | 1
sweating (General disorders) | 0 | 1 | 0 | 0
weakness (General disorders) | 0 | 0 | 0 | 2
aching of the intravenuos line (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
cavernoma left occipital cerebrum (Nervous system disorders) | 0 | 0 | 1 | 0
croakiness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
dry nose (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
flu-like symptoms (Infections and infestations) | 0 | 0 | 1 | 0
frequent dejection (Gastrointestinal disorders) | 0 | 1 | 0 | 0
gain of weight (General disorders) | 1 | 0 | 0 | 0
haemorrhagic cystitis (Renal and urinary disorders) | 0 | 1 | 0 | 0
hair loss (General disorders) | 0 | 0 | 0 | 1
hardening of arm/leg (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0
hearing loss (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
high gammaglobuline/alpha-1-globuline (Hepatobiliary disorders) | 0 | 0 | 1 | 0
high LDH (Hepatobiliary disorders) | 0 | 0 | 1 | 1
decubitus ulcer both ears (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
itching (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
pruritus at the eyelids (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
rash (Skin and subcutaneous tissue disorders) | 3 | 0 | 2 | 2
reddened hands (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
redness at puncture (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 5
redness of eyelid (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
redness on backside (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
swelling of arm/leg (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
aphtha (Gastrointestinal disorders) | 1 | 0 | 0 | 0
brown coated tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 1
coated tongue (Gastrointestinal disorders) | 0 | 1 | 0 | 0
constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
diarrhea (Gastrointestinal disorders) | 1 | 1 | 4 | 6
discomfort over the liver area (Gastrointestinal disorders) | 0 | 0 | 0 | 1
dry lips (Gastrointestinal disorders) | 0 | 1 | 0 | 0
dry mucosa mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 1
heartburn (Gastrointestinal disorders) | 1 | 0 | 0 | 0
inappetance (Gastrointestinal disorders) | 0 | 0 | 1 | 1
inappetence (Gastrointestinal disorders) | 0 | 1 | 0 | 0
mucositis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
nausea (Gastrointestinal disorders) | 2 | 3 | 1 | 5
obstipation (Gastrointestinal disorders) | 2 | 0 | 1 | 0
oral lesions due to dental prosthesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
pain during swallowing (Gastrointestinal disorders) | 1 | 0 | 0 | 0
red-brown coated tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 1
sialorrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
sore throat (Gastrointestinal disorders) | 0 | 0 | 2 | 0
swallow pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
vomiting (Gastrointestinal disorders) | 2 | 3 | 0 | 2
xerostomia (Gastrointestinal disorders) | 0 | 0 | 0 | 2
yellow coated tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 1
bleeding at puncture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 3
bleeding operation wound left shoulder (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
bloody sputum (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
haemoptysen (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
hematoma (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
hematoma at the neck (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
hematoma due to blood sampling (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
hematoma left arm (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
hemorrhoids bleeding (Gastrointestinal disorders) | 0 | 1 | 1 | 0
nosebleed (Blood and lymphatic system disorders) | 1 | 2 | 2 | 2
petechiae (Blood and lymphatic system disorders) | 2 | 0 | 4 | 2
red spots at the lower abdominal area (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
red spots, pustules (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
redness and bleeding of anus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
urinary bleeding (Renal and urinary disorders) | 0 | 1 | 0 | 0
elevated bilirubin (Hepatobiliary disorders) | 0 | 0 | 0 | 1
elevated liver test (alt) (Hepatobiliary disorders) | 0 | 0 | 0 | 1
high ALT (Hepatobiliary disorders) | 2 | 0 | 0 | 2
high AP (Hepatobiliary disorders) | 2 | 0 | 1 | 6
high AST (Hepatobiliary disorders) | 2 | 0 | 0 | 1
high billirubin (Hepatobiliary disorders) | 1 | 0 | 0 | 0
high direct bilirubin (Hepatobiliary disorders) | 0 | 0 | 0 | 1
high gGT (Hepatobiliary disorders) | 4 | 0 | 0 | 5
high GPT (Hepatobiliary disorders) | 2 | 0 | 0 | 0
high total bilirubin (Hepatobiliary disorders) | 0 | 0 | 0 | 1
hyperbilirubinemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1
intermittant elevated alt (Hepatobiliary disorders) | 0 | 0 | 0 | 1
low cholinesterase (Hepatobiliary disorders) | 0 | 0 | 0 | 1
low pancreas amylase (Hepatobiliary disorders) | 0 | 0 | 0 | 1
febrile neutropenia (Infections and infestations) | 0 | 0 | 1 | 0
fever (Infections and infestations) | 2 | 3 | 1 | 3
fever in neutropenia (Infections and infestations) | 1 | 0 | 0 | 0
herpes infection (Infections and infestations) | 0 | 0 | 0 | 1
herpes simplex infection lips (Infections and infestations) | 0 | 1 | 0 | 0
high procalcitonin (Infections and infestations) | 0 | 0 | 0 | 1
infection at the puncture of central ven (Infections and infestations) | 0 | 0 | 1 | 0
infection of puncture at central venous (Infections and infestations) | 0 | 0 | 1 | 0
infection with staphylococcus (Infections and infestations) | 0 | 0 | 3 | 0
infection with streptococcus mitis (Infections and infestations) | 0 | 0 | 1 | 0
klebsiella detection in sputum (Infections and infestations) | 0 | 0 | 0 | 1
rhinitis (Infections and infestations) | 1 | 0 | 0 | 0
swelling of the mucosa at the bottom of (Infections and infestations) | 0 | 0 | 1 | 0
thrombophlebitis (Infections and infestations) | 1 | 0 | 0 | 1
urethritis (Infections and infestations) | 0 | 0 | 0 | 1
urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 3
alkaline phophatase increase (Hepatobiliary disorders) | 0 | 0 | 0 | 1
elevated uric acid (Renal and urinary disorders) | 0 | 0 | 0 | 1
high creatinine (Renal and urinary disorders) | 1 | 0 | 0 | 2
high urea (Renal and urinary disorders) | 0 | 1 | 0 | 0
high uric acid (Renal and urinary disorders) | 0 | 0 | 1 | 0
hypalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
hypercalcelmia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
hyperchloridemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
hyperglykemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4
hyperkalemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 5
hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
hyperuricemia (Renal and urinary disorders) | 0 | 0 | 0 | 1
hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
hypocalcemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 5
hypokalemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 6
hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2
intermittant hypoalbuminia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
intermittent hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
low albumin (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
low albumine (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
low protein (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
calf cramps (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
swelling of arm/leg (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
amentia (Psychiatric disorders) | 0 | 1 | 0 | 0
confusion (Nervous system disorders) | 0 | 0 | 0 | 1
hallucination (Nervous system disorders) | 1 | 0 | 0 | 1
intermittant sleep disturbance (Nervous system disorders) | 1 | 0 | 0 | 0
intermittend sleeping disorder (Nervous system disorders) | 0 | 0 | 0 | 1
neuropathia aboth arms (Nervous system disorders) | 0 | 0 | 0 | 1
paraesthesia (fingers) (Nervous system disorders) | 0 | 0 | 0 | 1
paraesthesia (limbs, lips, fingers) (Nervous system disorders) | 0 | 0 | 0 | 1
patient not addressable (Nervous system disorders) | 0 | 0 | 0 | 1
prickle and numbness in both feet (Nervous system disorders) | 0 | 1 | 0 | 0
restlessness (Nervous system disorders) | 0 | 0 | 0 | 1
sleep disturbance (Nervous system disorders) | 1 | 0 | 0 | 0
slight drowsiness during caspofungin inf (Nervous system disorders) | 0 | 0 | 0 | 1
small pupils (Nervous system disorders) | 0 | 0 | 0 | 1
tremor (Nervous system disorders) | 0 | 0 | 0 | 1
viewing of colours (Nervous system disorders) | 0 | 0 | 1 | 0
worsening of visual acuity (Nervous system disorders) | 0 | 1 | 0 | 0
reddened eyes (Eye disorders) | 0 | 0 | 0 | 1
abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
ague (Infections and infestations) | 2 | 0 | 0 | 0
back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
backache (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
bonepain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
flank pain (General disorders) | 0 | 0 | 0 | 1
headache (Nervous system disorders) | 2 | 2 | 2 | 2
joint pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
kneepain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
muscle pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
neck aches (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
neck ache (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
neck pain (osteoporosis) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
neck stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
pain at puncture of the central venous c (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
pain at the costal arch (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
pain in the left arm (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
pain in thorax and abdomen (Gastrointestinal disorders) | 0 | 1 | 0 | 0
pain left calf (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
pain left upper arm (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
pain on central venous catheder punction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
pain stomach left site (General disorders) | 1 | 0 | 0 | 0
painful peripheral catheter punktion pla (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
painful shoulder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
pressure pain on the fingernails (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
slight backpain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
thoracic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
bronchospasms (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
cold (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 3
cough, bloody sputum (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0
hoarse voice (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
local pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
nasal discharge (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
pain int the lungs (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
pain while breathing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
patients feels like he has a common cold (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
worsening of breathing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
yellow expectoration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
acute renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
pollakisuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
polyuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
reduced urine production (Renal and urinary disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No